CLINICAL TRIAL: NCT02092376
Title: The Link Between Obesity And Vitamin D in Bariatric Patients With Omega-loop Bypass Surgery: a Randomized Controlled, Double-blinded Clinical Supplementation Trial
Brief Title: The Link Between Obesity And Vitamin D in Bariatric Patients With Omega-loop Bypass Surgery
Acronym: LOAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maria Luger (Other)
Responsible Party: Sponsor-Investigator, Maria Luger, Maria Luger, MSc, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LOAD; 2013-003546-16 (EudraCT Number)
Record Dates: First submitted 2014-03-17; First posted 2014-03-20 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Bariatric Surgery Candidate
Keywords: Bariatric surgery; vitamin D; supplementation
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): The loading dose of 300 000 IU is divided into three doses (100 000 IU) and will be given over the first months. All patients in the intervention group will receive the first loading dose of 100 000 IU at day of discharge. The second (2 weeks) and third (4 weeks postoperative) administration will be given based on the 25-hydroxy vitamin D concentration. After the last respectively third loading dose a maintenance dose of 3420 IU per day should maintain the high 25-hydroxy vitamin D concentration. It should be administered for up to 46 weeks (until follow-up visit)
  Interventions: Drug: Cholecalciferol
- Placebo (Placebo Comparator): The placebo loading dose (oil) is divided into three administrations and will be given over the first months. All patients in the placebo group will receive the first placebo loading dose at day of discharge. After the last placebo loading dose a maintenance dose of 3420 IU per day should maintain the 25-hydroxy vitamin D concentration. It should be administered for up to 46 weeks (until follow-up).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cholecalciferol
  Arms: Intervention
Drug: Placebo
  Arms: Placebo

SUMMARY:
The aim of the study is to increase vitamin D concentrations or to keep it on high level, respectively, by supplementing with vitamin D3 in a different dose regime, and to improve the overall health status in bariatric patients. In this project, the vitamin D status, the parameters of inflammation, bone turnover, insulin resistance, liver and depression score of bariatric patients are expected to improve, due to supplementation of a loading dose compared to the standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Planned omega loop bypass surgery
* 25-hydroxy vitamin D < 75 nmol/l
* BMI >40 or ≥35 kg/m2 with co-morbidities e.g. diabetes mellitus, hypertension
* Body weight <140 kg (due to limitation of DEXA measurement)
* Capability to consent

Exclusion Criteria:

* Another planned form of bariatric surgery
* Hypercalcemia (calcium >2.63 mmol/l) or hypocalcemia (<1.75 mmol/l)
* Renal insufficiency (creatinine >133 μmol/l or GFR <50 ml/min)
* Primary hyperparathyroidism
* Malignancy
* Infection e.g. human immunodeficiency virus
* Medical conditions requiring daily calcium supplements or antacid use
* Known hypersensitivity to cholecalciferol
* No capability to consent
* Imprisoned persons

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
25-hydroxy vitamin D levels | 24 weeks postoperatively
  25-hydroxy vitamin D levels after 24 weeks measured in intervention and placebo group, adjusting for the baseline value as covariate

SECONDARY OUTCOMES:
Prevalence of sufficient vitamin D | 24 weeks postoperatively
  Number of patients reaching 25-hydroxyvitamin D levels above 75 nmol/l
Prevalence of vitamin D deficiency | 24 weeks postoperatively
  Prevalence of vitamin D deficiency
Co-morbidities | 24 weeks postoperatively
  Prevalence of Co-morbidities
Prescribed medication | 24 weeks postoperatively
  Change in prescribed medication
Body weight, body composition | 24 weeks postoperatively
  Change in body weight and body composition by bioelectrical impedance analysis
Blood pressure | 24 weeks postoperatively
  Change of vital signs (blood pressure)
Laboratory parameters | 24 weeks postoperatively
  Change in laboratory parameters compared to baseline: vitamin D status, bone turnover markers, calcium homeostasis, parathyroid hormone, inflammation, insulin resistance
Depression symptoms | 24 weeks postoperatively
  Prevalence of depression symptoms assessed by Beck Depression Inventory Questionnaire
Bone mineral density and body fat content | 24 weeks postoperatively
  Assessment of bone mineral density and total body fat content by DEXA
Liver condition | 24 weeks postoperatively
  Measurement of liver stiffness and fat content by FibroScan and CAP
Dietary assessment | 24 weeks postoperatively
  Dietary assessment will be documented with a 5-day food record to calculate vitamin D intake and the Mediterranean Score (questionnaire with calculated score)
Gut microbiota composition | 24 weeks postoperatively
  Association between vitamin D, gut microbiota and surgery-induced weight loss, by collecting stool samples
Vitamin D in adipose and liver tissue | during surgery
  For instance, for the purposes of describing adipose depot vitamin D concentrations and expression of enzymes in subcutaneous, visceral adipose and liver tissue samples will be collected during the omega loop gastric bypass surgery. Furthermore, the liver tissue samples should be used in addition for a histological examination as extended diagnostics (NAFLD/ NASH).

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Ludvik, M.D., Principal Investigator — Division of Endocrinology & Metabolism, Department of Internal Medicine III, Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Chakhtoura MT, Nakhoul NF, Akl EA, Safadi BY, Mantzoros CS, Metzendorf MI, El-Hajj Fuleihan G. Oral vitamin D supplementation for adults with obesity undergoing bariatric surgery. Cochrane Database Syst Rev. 2024 Oct 1;10(10):CD011800. doi: 10.1002/14651858.CD011800.pub2. PMID 39351881
- [Derived] Kruschitz R, Wakolbinger M, Schindler K, Prager G, Hoppichler F, Marculescu R, Ludvik B. Effect of one-anastomosis gastric bypass on cardiovascular risk factors in patients with vitamin D deficiency and morbid obesity: A secondary analysis. Nutr Metab Cardiovasc Dis. 2020 Nov 27;30(12):2379-2388. doi: 10.1016/j.numecd.2020.08.011. Epub 2020 Aug 20. PMID 32981799
- [Derived] Luger M, Kruschitz R, Winzer E, Schindler K, Grabovac I, Kainberger F, Krebs M, Hoppichler F, Langer F, Prager G, Marculescu R, Ludvik B. Changes in Bone Mineral Density Following Weight Loss Induced by One-Anastomosis Gastric Bypass in Patients with Vitamin D Supplementation. Obes Surg. 2018 Nov;28(11):3454-3465. doi: 10.1007/s11695-018-3353-2. PMID 29968187
- [Derived] Luger M, Kruschitz R, Kienbacher C, Traussnigg S, Langer FB, Prager G, Schindler K, Kallay E, Hoppichler F, Trauner M, Krebs M, Marculescu R, Ludvik B. Vitamin D3 Loading Is Superior to Conventional Supplementation After Weight Loss Surgery in Vitamin D-Deficient Morbidly Obese Patients: a Double-Blind Randomized Placebo-Controlled Trial. Obes Surg. 2017 May;27(5):1196-1207. doi: 10.1007/s11695-016-2437-0. PMID 27837387
- [Derived] Luger M, Kruschitz R, Kienbacher C, Traussnigg S, Langer FB, Schindler K, Wurger T, Wrba F, Trauner M, Prager G, Ludvik B. Prevalence of Liver Fibrosis and its Association with Non-invasive Fibrosis and Metabolic Markers in Morbidly Obese Patients with Vitamin D Deficiency. Obes Surg. 2016 Oct;26(10):2425-32. doi: 10.1007/s11695-016-2123-2. PMID 26989059
- [Derived] Luger M, Kruschitz R, Marculescu R, Haslacher H, Hoppichler F, Kallay E, Kienbacher C, Klammer C, Kral M, Langer F, Luger E, Prager G, Trauner M, Traussnigg S, Wurger T, Schindler K, Ludvik B. The link between obesity and vitamin D in bariatric patients with omega-loop gastric bypass surgery - a vitamin D supplementation trial to compare the efficacy of postoperative cholecalciferol loading (LOAD): study protocol for a randomized controlled trial. Trials. 2015 Aug 5;16:328. doi: 10.1186/s13063-015-0877-9. PMID 26242295